CLINICAL TRIAL: NCT03787992
Title: A Randomized, Double-blind, Positive-controlled, Multi-center Phase III Clinical Study of Evaluating Alflutinib Mesylate Versus Gefitinib as First-line Therapy in Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC) With EGFR-sensitive Mutations（FlAG）
Brief Title: Alflutinib Mesylate Versus Gefitinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer （FLAG）
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201801215
Record Dates: First submitted 2018-12-18; First posted 2018-12-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced or Metastatic EGFR Sensitising Mutation Positive Non-small Cell Lung Cancer
MeSH Terms: interventions — aflutinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alflutinib Mesylate (AST2818) +placebo (Experimental): AST2818 (80 mg or 40 mg orally, once daily) plus placebo Gefitinib (250 mg orally, once daily), in accordance with the randomization schedule
  Interventions: Drug: Alflutinib Mesylate (AST2818) 80mg//40 mg+ placebo; Drug: Placebo Gefitinib 250 mg
- Gefitinib + placebo AST2818 (Active Comparator): Gefitinib (250 mg orally, once daily) + placebo AST2818 (80 mg or 40 mg orally, once daily), in accordance with the randomisation schedule.
  Interventions: Drug: Gefitinib 250 mg; Drug: Placebo AST2818 80mg//40 mg

INTERVENTIONS:
Drug: Alflutinib Mesylate (AST2818) 80mg//40 mg+ placebo — The initial dose of AST2818 80 mg once daily can be reduced to 40 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Alflutinib Mesylate (AST2818) +placebo
Drug: Placebo Gefitinib 250 mg — The initial dose of Placebo Gefitinib 250 mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Alflutinib Mesylate (AST2818) +placebo
Drug: Gefitinib 250 mg — The initial dose of Gefitinib 250mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Gefitinib + placebo AST2818
Drug: Placebo AST2818 80mg//40 mg — The initial dose of Placebo AST2818 80 mg once daily can be reduced to Placebo AST2818 40 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Gefitinib + placebo AST2818

SUMMARY:
To assess the efficacy and safety of Alflutinib Mesylate versus Gefitinib in patients with locally advanced or Metastatic Non Small Cell Lung Cancer

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomised study assessing the efficacy and safety of Alflutinib Mesylate (AST2818) (80 mg orally, once daily) versus Gefitinib (250 mg orally, once daily] in patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) that is known to be EGFR sensitising mutation (EGFRm) positive for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet all the following criteria to be enrolled in this study: subjects will voluntarily participate and sign a written informed consent.
2. Male or female, aged at least 18 years.
3. ECOG performance status of 0 to 2. Life expectancy of at least 12 weeks.
4. Patients had histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma not amenable to curative surgery or radiotherapy.
5. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R).
6. Tumour tissue sample in a quantity sufficient to allow for central analysis of EGFR mutation status.
7. Patients must be treatment-naïve for locally advanced or metastatic NSCLC and eligible to receive first-line treatment with gefitinib or erlotinib as selected by the participating centre. Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) if the disease has no progression during one year.
8. At least one measurable lesion by CT or MRI. The measureable lesion should receive no local treatments (i.e., radiotherapy) or not used for screening biopsies (If there is only one target lesion that must be biopsied, baseline tumor evaluation is required at least 14 days after screening biopsy) and can be accurately measured at baseline with the longest diameter greater than 10 mm at baseline (if it is a lymph node, short diameter greater than 15 mm is required). If the lesions located at the regions which were previously treated are confirmed to progress, they can be chosen as lesion according to RECIST Version 1.1
9. Females who have fertility potential before menopause should have a pregnancy test in the time period of 7 days prior to start of dosing, should not be breast feeding and must have a negative pregnancy test (blood test or urinalysis) prior to start of dosing; Males and females of child-bearing age must take adequate contraceptive measures within 3 months after signing the informed consent of the study to the last drug treatment.

Exclusion Criteria:

1. Treatment with any of the following:

   * Prior treatment with any systemic anti-cancer therapy for locally advanced/metastatic NSCLC, such as standard chemotherapy, targeted therapy, biological therapy, immune therapy and for the prior adjuvant / neo-adjuvant therapy listed in the inclusion criteria VII
   * Patients received other systemic anticancer therapies for advanced/metastatic non-small cell lung cancer
   * Patients who have received intrapleural perfusion therapy should be admitted to the group unless the stabilization of hydrothorax is longer than 28 days
   * Prior treatment with an EGFR-TKI
   * Major surgery within 4 weeks of the first dose of study drug
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug and local radiotherapy or palliative radiotherapy for bone metastasis within 14 days before first drug administration
   * Patients receiving medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP) 3A4 within 7 days before first drug administration and patients continuously taking these medications during investigating period
   * Patients taking traditional Chinese medicine and preparations whose therapeutic goal is anti-tumors within 7 days before first drug administration; or continuously taking these medications during investigating period
   * Patients with any factors that increase the risk of QTc prolongation or risk of Torsade ventricular tachycardia event who continuously take these medications during investigating period.
   * Before the first administration, the duration of discontinuation of other clinical experimental drugs was less than 14 days
2. Unrecovered toxic reaction due to anti-tumor therapy existed, with over 1 grade of CTCAE (except alopecia) or 2 grade if ever applied DDP curing related neuropathy; Bone marrow, liver and kidney organ function please refer to exclusion criteria 7.
3. The tissue type is mixed type, that is, patients with lung adenocarcinoma mixed with lung squamous cell carcinoma.
4. Patients with spinal cord compression, asymptomatic and stable brain metastases, except for those patients who have completion of the definitive therapy and steroids at least 28 days before investigation，or patients who received local radiotherapy for brain metastasis will be allowed in when the period of stabilization of brain metastases are at no shorter than 28 days.
5. Patients with other malignant tumors or have a history of other malignant tumors, except for basal cell carcinoma of the skin, carcinoma in situ of the cervix and ductal carcinoma in situ of the breast.
6. Any condition affecting the drug taking, or significantly affecting the absorption or the pharmacokinetic parameters, include any kind of uncontrollable nausea or vomit, chronic gastroenteropathy, disability in swallowing, history of gastrointestinal resection or surgery, uncured recurrent diarrhea, atrophic gastritis (the age of onset is less than 60 years old), stomach diseases, crohn's disease and ulcerative colitis that require long-term use of PPI antiacid drugs without cure.
7. Patients of organ insufficiency in bone marrow, liver and kidney meet the following requirements (patients should receive no blood transfusion, blood product, hematopoietic stimulating factors, and albumin two weeks before blood sampling of admission )：

   * Absolute neutrophil count < 1.5 x 109/L, Platelet count < 75 x109/L, Haemoglobin < 90 g/L;
   * Alanine aminotransferase/Aspartate aminotransferase > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times in the presence of liver metastases;
   * Total bilirubin > 1.5 times ULN, or >3 times ULN in the presence of definitive Gilbert's syndrome (Unbound hyperbilirubinemia) or liver metastases;
   * Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated by Cockcroft and Gault equation);
   * The international standardized ratio (INR) was > and 1.5, and the partial activation time of prothrombin (APTT) was > 1.5 times ULN.
8. Any condition meets the following cardiac standard:

   * Mean resting corrected QT interval (QTc)>470 msec, obtained from 3 ECG, using the screening clinic ECG machine-derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
   * Echocardiographic examination: LVEF<50%
9. Active infection with HBV, HCV, or HIV. All subjects will be screened for HBV, HCV, or Or HIV infection during the screening period:

   * HBsAg positive, HBV DNA ≥1000cps/ml（or200IU/ml）
   * Anti-HCV antibody was positive and HCV RNA was positive
   * HIV antibody was positive
10. Interstitial lung disease, drug - induced interstitial pulmonary disease, history of radiation pneumonia which required steroid treatment; acute or progressive pulmonary symptoms may occur at baseline or interstitial pulmonary disease may be identified that the researchers considered not suitable for trail
11. Allergy to the study drug and/or its excipients is known or suspected
12. Women during pregnancy or lactation
13. Judgment by investigator that the patients should participate in the study if the patient is unlikely to comply with study procedure, restrictions, and requirements (for example, uncontrolled hypertension, uncontrolled diabetes, active bleeding constitution, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) (Months) | At baseline and every 6 weeks for the first 17 months and then every 12 weeks relative to randomisation until progression ( (approximately 12 months)
  Progression-free survival was defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression and was used to assess the efficacy of single agent alflutinib compared with SoC EGFR-TKI therapy as measured by PFS.

SECONDARY OUTCOMES:
Overall Survival (OS)- Number of Participants With an Event | From first dose to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks (approximately 29 months)
  Overall survival was defined as the time from the date of randomisation until death from any cause and was used to further assess the efficacy of alflutinib compared with SoC EGFR-TKI therapy
Progression Free Survival (PFS) evaluated by investigator | At baseline and every 6 weeks for the first 17 months and then every 12 weeks relative to randomisation until progression (approximately 12 months)
  Progression-free survival was defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression and was used to assess the efficacy of single agent alflutinib compared with SoC EGFR-TKI therapy as measured by PFS.
Objective Response Rate (ORR) | At baseline and every 6 weeks for the first 17 months and then every 12 weeks relative to randomisation until progression (approximately 12 months)
  ORR was defined as the number (%) of patients with measurable disease with at least 1 visit response of Complete response (CR) or Partial response (PR) and it was used to further assess the efficacy of alflutinib compared with SoC EGFR-TKI therapy
Duration of Response (DoR) | At baseline and every 6 weeks for the first 17 months and then every 12 weeks relative to randomisation until progression (approximately 12 months)
  Duration of response was defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression and was used to further assess the efficacy of alflutinib compared with SoC EGFR-TKI therapy.
Depth of Response | At baseline and every 6 weeks for the first 17 months and then every 12 weeks relative to randomisation until progression (approximately 12 months)
  The Depth of response was defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions (TLs) at the nadir, in the absence of new lesions (NLs) or progression of Non-target lesions (NTLs), compared to baseline and was used to further assess the efficacy of alflutinib compared with SoC EGFR-TKI therapy
Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) Questionnaires Lung Cancer 13 (QLQ-LC13) | Questionnaires completed at week 1, 4, 7, 9, 12, 15 , 18,21,27,33,39,45and51
  The EORTC QLQ-LC13 was a lung-cancer-specific module comprising 13 questions to assess lung cancer symptoms (cough, haemoptysis, dyspnoea, and site-specific pain [pain in chest, pain in arm or shoulder, and pain in other parts); treatment related side-effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia); and pain medication. Except for a multi-item scale for dyspnoea, all were single items. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items. Higher scores on the global health status/QoL and functioning scales indicated better health status/QoL and better function. Higher scores on the symptoms scales indicated greater symptom burden. The results of the analyses were presented in terms of a least squares mean together with its associated 95% profile likelihood CI
Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items | Questionnaires completed at week 1, 4, 7, 9, 12, 15 , 18,21,27,33,39,45and51
  he EORTC QLQ-C30 cancer-specific questionnaire consisted of 30 questions, which were combined to produce 5 functional scales (Physical, Role, Cognitive, Emotional, Social); 3 symptom scales (Fatigue, Pain, Nausea/Vomiting); 6 individual items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties); and a global measure of health status/QoL. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, the functional scales, and the global health status/QoL scale in the EORTC QLQ-C30. Higher scores on the global health status and functioning scales indicated better health status/function. Higher scores on the symptoms scales indicated greater symptom burden. The results of the analyses were presented in terms of a least squares mean together with its associated 95% profile likelihood CI.

CONTACTS AND LOCATIONS:
Locations (1):
- cancer hospital Chinese academy of medical sciences, Beijing, China

REFERENCES:
- [Derived] Shi Y, Chen G, Wang X, Liu Y, Wu L, Hao Y, Liu C, Zhu S, Zhang X, Li Y, Liu J, Cao L, Cheng Y, Zhao H, Zhang S, Zang A, Cui J, Feng J, Yang N, Liu F, Jiang Y, Gu C; FURLONG investigators. Furmonertinib (AST2818) versus gefitinib as first-line therapy for Chinese patients with locally advanced or metastatic EGFR mutation-positive non-small-cell lung cancer (FURLONG): a multicentre, double-blind, randomised phase 3 study. Lancet Respir Med. 2022 Nov;10(11):1019-1028. doi: 10.1016/S2213-2600(22)00168-0. Epub 2022 Jun 2. PMID 35662408